CLINICAL TRIAL: NCT00959309
Title: Media Use in Preschooler Study (MUPS) An Office Based Intervention to Improve Media Use in Preschool Children: a Randomized Controlled Trial
Brief Title: Media Use in Preschooler Study (MUPS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Catherine Birken, Staff Paediatrician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1000009542
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Obesity
Keywords: pediatrics; media; MUPS
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Strategies to decrease screen time in children
- Control (Active Comparator)
  Interventions: Behavioral: Non-Strategical Media Education

INTERVENTIONS:
Behavioral: Strategies to decrease screen time in children — 15 minute session about the health impact of screen time in children and strategies to decrease screen time (removing televisions from the child's bedroom, budgeting screen time, providing a contingency plan for time spent not watching TV, encouraging family meal time, and implementing a one week television turn off, where children are encouraged to spend one week without watching TV/videos). Activities for the child include reading a story about television viewing (The Berenstain Bears and Too Much TV), and creating a list of non TV related activities to replace TV time. The intervention group will receive a CPS handout titled 'Promoting Good Television Habits' and a calendar with stickers for the television turn off.
  Educational session on good media use (information on television rating systems, internet safety, and limiting exposure to violent programming, and the CPS handout entitled 'Managing Media in the Home')
  Arms: Intervention
Behavioral: Non-Strategical Media Education — Educational session on good media use (information on television rating systems, internet safety, and limiting exposure to violent programming, and the CPS handout entitled 'Managing Media in the Home')
  Arms: Control

SUMMARY:
Childhood obesity is an epidemic and increasing. There are very few effective treatments for obesity in children. Recent studies have shown an association between obesity and sedentary behaviors such as television, video viewing and playing video games ('screen time') in preschool aged children. A school based intervention to reduce screen time in older children has been effective in preventing obesity.

The reduction of screen time may lead to the prevention of obesity and its complications in preschool children.

DETAILED DESCRIPTION:
There have been no trials examining an intervention to decrease screen time in preschool children in the physician office setting. This setting is appealing for interventions directed to preschool children because of accessibility. In addition, other public health interventions implemented in a physician office setting, such as home safety advice, have been effective.

The proposed study design will be a randomized controlled trial. The intervention group will receive the study intervention, which is a 15 minute session about the health impact of screen time in children and strategies to decrease screen time.

The objective of this study is to determine if an office based intervention is effective in decreasing screen time (television, video viewing and playing video games) in preschool children.

ELIGIBILITY:
Inclusion Criteria:

* registered to attend a 3 year old well child visit

Exclusion Criteria:

* children with limitations in ambulation or cognitive delay will be excluded from the study.

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Parent reported number of hours screen time on the previous weekday and previous weekend day | 6 and 12 months

SECONDARY OUTCOMES:
Number of meals in front of the TV | 6 and 12 months
Activity levels | 6 and 12 months
Anthropometric measures | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Birken, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada